CLINICAL TRIAL: NCT03694769
Title: Developing a Psychological Understanding of Idiopathic Drop Attacks
Brief Title: Investigating Drop Attacks
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Emily Revell, Trainee Clinical Psychologist, University of Edinburgh
Other Study IDs: CAHSS1710/03
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Functional Disorder
Keywords: functional neurological symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: Semi-structured interview and drop attack diary
  Interventions: Other: Semi-structured interview; Other: Drop attack diary

INTERVENTIONS:
Other: Semi-structured interview — One-hour interview with researcher
Other: Drop attack diary — Diary of any drop attacks experienced within an 8 week period

SUMMARY:
The aim of this project is to better understand the experiences of people who have idiopathic drop attacks. These falls have no identified medical cause but can cause people injuries such as bruising, facial injuries and, in some cases, broken bones. It can also make them worry about having more falls, and the pain and embarrassment this would cause, and stop them from going out. There has been very little research in this area and there are currently no treatments.

In this study, ten people who experience idiopathic drop attacks will be interviewed at an outpatient clinic to understand more about them and the falls. They will be asked in particular about the period of time around when they started having the falls and whether there are aware of any triggers. Participants will also be asked to write accounts of these drop attacks, after they have happened, for a period of eight weeks. They will be asked to describe what they were thinking and feeling, and how they felt in themselves before and after the fall.

This information will allow the researcher to look at common experiences that people who experience these falls have. This understanding could help to identify whether a psychological approach to treatment could help individuals to manage and cope with this condition.

DETAILED DESCRIPTION:
Design

In this exploratory qualitative study, neurology outpatients with ongoing Idiopathic Drop Attacks (IDAs) will undergo psychological assessment and complete written diaries for eight weeks. Throughout the study, participants will receive treatment as usual from a neurologist.

Procedure

Participants will be recruited from a neurology outpatient clinic at the Department of Clinical Neurosciences in Edinburgh where they will be approached by their consultant who will give them a participant information sheet. If they are interested in taking part, a meeting will be set up with the researcher to discuss the study further and obtain written informed consent.

Participants will then meet with the researcher to complete an initial psychological interview which will be audio recorded. This interview will follow a standard initial psychological interview structure and will aim to gain information about the person's experiences of IDAs, along with relevant personal and social history.

Following this initial interview, participants will be asked to record written accounts of any IDA, detailing their thoughts, physical arousal, feelings and behaviour, as close to the event as possible. They will be encouraged to record detailed accounts, outlining the period before, during and after the episode, in order to identify any potential triggers. They will be shown an example of a completed diary in order to help them to understand what they need to do. Participants will be asked to record such events over a period of eight weeks during which the researcher will contact them fortnightly to discuss any difficulties or concerns. If participants do not experience any drop attacks during this period, they will be asked if they want to continue recording diaries for an additional two to four weeks.

Following completion of this period, participants will meet again with the researcher to return the diaries and discuss any patterns noticed in the interview and diaries. The researcher will also answer any further questions that the participant has about the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18+
2. Idiopathic drop attacks occurring 6+ times per year
3. Having previously completed extensive investigation into possible cause of drop attacks
4. Able to provide informed consent

Exclusion Criteria:

1. Diagnosis which would provide an alternative explanation for drop attacks
2. Drop attacks due to malfunction of the lower limbs, changes in body or head posture, or vertigo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a single functional neurological disorders clinic at the Western General Hospital in Edinburgh.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Semi-structured assessment interview | One hour
  This audio-recorded 60-minute interview will follow the format of an initial psychological assessment and will allow discussion of presenting problems and relevant personal and social history. This will allow potential predisposing and precipitating factors to be identified. Participants' experiences of IDAs will also be discussed, focussing on thoughts, feelings and behaviour before and after the episodes. The participants will also be asked about the impact that these have had on their everyday functioning.

SECONDARY OUTCOMES:
Drop attack diary | 8 weeks
  Participants will be asked to write an account of any IDAs. They will be shown an example diary and will also be given a prompt sheet, asking them to recall any triggers, feelings, physical arousal, thoughts and behaviour both directly before and after the episode. This diary will be completed by participants as close to the episode as possible

CONTACTS AND LOCATIONS:
Locations (1):
- Western General Hospital (NHS Lothian), Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All anonymised research data will be stored for 10 years by the University of Edinburgh, in line with MRC requirements. Identifiable information with not be shared with other researchers, and will be destroyed within six months of the study ending.

DOCUMENTS (1):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03694769/Prot_000.pdf